CLINICAL TRIAL: NCT07014969
Title: En-bloc Versus Lobe-by-lobe Holmium Laser Enucleation of the Prostate (HoLEP): A Randomized Controlled Trial
Brief Title: En-bloc With Early Apical Release Versus Lobe-by-lobe LASER Enucleation of the Prostate
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Yahya Hossam, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.21.07.1561
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostate Hyperplasia; Bladder Outlet Obstruction
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder Neck Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- En-bloc HoLEP (Experimental): 1. An inverted U-shaped incision in front of the veru montanum followed by extension of the incision laterally on both lateral lobes
  2. Using the peak of the scope, blunt enucleation of the lateral lobes
  3. Enucleation continued laterally with insinuation of the scope lateral to the enucleated lobe on both sides, ending by residual mucosal attachment of the adenoma to the sphincter between 11 and 1 O'clock positions
  4. Release of the adenoma from the sphincter is done by transverse cutting of the mucosal attachment using 180 degree inverted scope the fiber position at 12 O'clock position of the scope
  5. the enucleation process continued above the adenoma from side to side both bluntly and laser assisted till reaching the bladder neck
  6. lateral dissection of the ad enoma will be carried out on both sides
  7. Finally basal dissection of the adenoma and flipping of the both adenomas as one chunk to the bladder followed by laser cutting of any residual attachment.
  Interventions: Procedure: En-bloc HoLEP
- Lobe by Lobe HoLEP (Active Comparator): classic 2 or 3 lobe technique with early apical release
  Interventions: Procedure: En-bloc HoLEP

INTERVENTIONS:
Procedure: En-bloc HoLEP — Removal of the whole adenoma in one piece using laser energy

SUMMARY:
Since its introduction in 1998 , and through numerous level 1a evidence, Holmium Laser enucleation of the prostate (HoLEP) has come to be considered a size-independent golden standard treatment for management of bladder outlet obstruction (BOO) secondary to benign prostatic hyperplasia (BPH) endorse by all guidelines.

Furthermore, Holep, together with minimaly invasive simple prostatectomy, is considered the most accepted alternative to Open simple protatectomy for prostates larger than 80ml.

Despite being the most thoroughly investigated laser technique with enduring efficacy and low morbidity, HoLEP remains restricted to relatively few centers mostly due to the long flat learning curve and lack of access to mentorship programs . On the other hand, the prevalence of stress urinary incontinence following HoLEP was reported to be about (3.3%-26% ) To overcome these difficulties hindering the wide-spread adoption of HoLEP, several modifications of the original three-lobe technique have been described to improve surgical outcomes and overcome the learning difficulties .

One of the newer modifications for AEEP that have shown promising results is the en-bloc enucleation with early apical release developed by Sancha et al in 2015 utilizing Green Light LASER which has the potential advantage of preserving the integrity of the external sphincter . The same principles of early apical liberation and sphincter mucosal preservation have been applied to lobe by lobe techniques as well.

In this work the investigators aim to obtain high level evidence of efficacy of En-bloc HoLEP and its impact on early recovery of continence in comparison to the conventional lobe-by-lobe (LBL) HoLEP.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is one of the most commonly diagnosed conditions of the male genitourinary tract worldwide, resulting in approximately 1.2 million surgical procedures per year. Holmium laser enucleation of the prostate (HoLEP) has proven to be an efficient, durable, and safe surgical option for the management of BPH. The European Association of Urology (EAU) Guidelines on Management of Non-Neurogenic Male Lower Urinary Tract Symptoms (LUTS) in 2016 considered HoLEP (referred to as endoscopic enucleation of the prostate, EEP) as a reference technique for the management of large prostates.

The evolution of laser technology has revived the concept of anatomical enucleation, allowing the resectoscope to be used to dissect the adenoma from the surgical capsule, mimicking the surgeon's index finger in open prostatectomy. This concept of laser-assisted anatomical enucleation can be efficiently replicated by other types of laser energy apart from Holmium.

HoLEP was first described in 1998 as a three-lobe technique, involving the creation of two incisions at the bladder neck, then joining these incisions in front of the verumontanum before enucleating the median, left, and right lobes sequentially but its dissemination has been limited by a steep learning curve and relative procedural difficulty, especially in large glands as well as high rate of trasnient stress urinary incontinence.

More recently, 'en bloc' techniques have been introduced, which may offer advantages such as better visualization, faster identification of the surgical capsule and dissection plane, early release and better preservation of the sphincter, and an improved learning curve compared to the three-lobe technique.

One such en-bloc method involves identifying the correct plane between adenoma and capsule at the apex of the left lobe lateral to the verumontanum, extending the incision retrogradely towards the bladder, and using the endoscope to gently raise the lobe from the capsular plane, gradually exposing the dissection plane and reducing intraoperative difficulties such as bleeding and capsule perforation, while shortening enucleation time.

Feasibility studies of en-bloc HoLEP on patients with moderately enlarged prostates showed promising operative times and significant reductions in prostate-specific antigen (PSA) and transition zone volume, indicating effective adenoma removal.

Comparative studies between en-bloc HoLEP and traditional two- or three-lobe techniques have reported shorter enucleation times and lower laser energy use with the en-bloc approach.

Large randomized trials have similarly found that en-bloc HoLEP is associated with significantly shorter operative and enucleation times compared to the three-lobe technique.

Aim of the work

Growing evidence suggests that en-bloc enucleation of the prostatic adenoma, which involves dissection of the adenoma as a single tissue mass, offers advantages over the usual two- or three-lobe techniques: shortened operation time, optimal visualization of the dissection plane due to reduced bleeding and excellent irrigation, and improved enucleation effectiveness.

Early demarcation of the 'white line' leading to early release of the sphincter from the prostatic apex could reduce the likelihood of transient postoperative stress urinary incontinence. This is because the sphincter is less likely to be stretched during dissection movements, which can otherwise occur when the external sphincter is fixed on one side and the scope is dissecting on the opposite side.

In this study, the investigators aim to provide high-level evidence on the feasibility and efficacy of en-bloc enucleation using holmium lasers and its impact on early continence recovery. The investigators will conduct a well-designed randomized controlled trial comparing en-bloc endoscopic laser enucleation versus the conventional two- or three-lobe technique.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age ≥ 40 years
2. LUTS secondary to BOO due to BPH who failed medical treatment
3. International prostate symptom scores (IPSS) >15 and bother score (QOL) ≥ 3 (according to IPSS question 8)
4. Peak urinary flow rate (Qmax) <15 ml/sec with at least 125 ml voided volume or Patients with acute urine retention secondary to BPH who failed trial of voiding on medical treatment.
5. ASA (American society of anaesthesiologists) score ≤3.
6. TRUS prostate size 80-200 ml

Exclusion Criteria:

1. Patient with neurological disorder which might affect bladder function as cerebrovascular stroke, Parkinson disease
2. Active urinary tract infection,
3. Presence of active bladder cancer.
4. Known prostate cancer patients will be excluded preoperatively on the basis of digital rectal examination, prostate specific antigen level, and TRUS imaging followed by prostate biopsies if necessary.
5. Patient has a disorder of the coagulation cascade (e.g., liver cell failure) or disorders that affect platelet count or function (e.g., von Willebrand disease) that would put the subject at risk for intraoperative or postoperative bleeding.
6. Patient is unable to discontinue anticoagulant and antiplatelet therapy preoperatively (3-5 d) except for low-dose aspirin (e.g., 100 mg).
7. Patient has had an acute myocardial infarction or open-heart surgery <180 days prior to the date of informed consent. -

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Enucleation efficiency | perioperative/ periprocedural
  resected prostate weight divided by enucleation time
enucleation speed | perioperative/ periprocedural
  time between insertion. of laser fiber till complete detachment of the adenoma

SECONDARY OUTCOMES:
Resected prostate weight | perioperative/ periprocedural
  Weight of resected prostatic tissue expressed in Grams
Incidence of early urinary incontinence | 1,3 and 6 months
  assessment of incidence of early urge and stress urinary incontinence.
morcellation efficiency | perioperative/ periprocedural
  Weight of resected prostate tissue in grams morcellated per minute expressed in (grams per minute)
length of hospital stay | perioperative/ periprocedural
  lenght of hospital admission measure in days
total laser energy | perioperative/ periprocedural
  Total Laser energy required expressed in Joules
LASER/Prostate ratio | perioperative/ periprocedural
  Laser energy required to resect one gram of prostatic tissue expressed in (kiloJoule per gram)
volume of intraoperative irrigation | perioperative/ periprocedural
  volume of irrigation saline volume expressed in Litres
perioperative blood loss | perioperative/ periprocedural
  haemoglobin deficit measured by the difference between preopeartive and postoperative hemoglobin expressed in Gm/dl
catheterization time | perioperative/ periprocedural
  time to catheter removal expressed in Days

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-Assmy, Study Director — Mansoura Univeristy
Locations (1):
- Urology and nephrology center, Al Mansurah, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No